CLINICAL TRIAL: NCT04834466
Title: Factors Associated With Pain Level Experience in Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chia Jung Lee (Other)
Collaborators: Shen Gaang Jong Shiaw Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Chia Jung Lee, Principal investigator, Alfonso X El Sabio University
Organization: Alfonso X El Sabio University (Other)
Other Study IDs: AlfonsoXElSabioU
Record Dates: First submitted 2021-03-19; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Orthodontic Pain; Pain; Orthodontic Appliance Complication
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pain Level experience during orthodontic treatment — A questionnaire was given to patients who have started their orthodontic treatment to assess their pain level experience

SUMMARY:
Orthodontic pain has been the primary concern from all patients who requires orthodontic treatment. The design of the study will help us comprehend how patient experienced and managed pain during their orthodontic treatment, average pain level in different orthodontic appliances and factors that could affect pain level experience during treatment, including gender, age, brackets types, hygiene level and habitude.

DETAILED DESCRIPTION:
To interpret the average pain level experience in orthodontic treatment and find correlations of different pain level within each individual from the clinical reports and questionnaires collected from each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient with orthodontic treatment over 2 months and less than 12 months
* Patient with braces or Invisalign
* Patient who goes to orthodontic visits routinely

Exclusion Criteria:

* Patient undergoing orthopaedic treatment (Functional appliances, 2x4 braces placement, maxillary expansion)
* Patient who do not understand Spanish
* Patient with cognitive impairment
* Patient who do not want to participate in the study
* Patient who have complete their orthodontic treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Clinic Centro Odontologo Innovaccion y especialidad avanzadas who are undergoing orthodontic treatment were selected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain level difference within different orthodontic appliances | From date of randomisation until the date of a 150 participation. Through study completion, an average of 1 year
  Orthodontic appliances such as Invisalign, conventional braces and self-ligated braces are included to compare. Pain assessed through visual analogue scale (VAS) rating 0(No pain) to 10(extreme pain) were given individually to participant with different orthodontic appliances to gather information. The lower the score, the lesser the pain and vise versa.

SECONDARY OUTCOMES:
Pain level difference within different factors | Through study completion, an average of 1 year.
  Factors such as gender, age, hygiene level, tooth discrepancies, habitude and mental state could affect the pain level experience during orthodontic treatment. Survey given with respective questions and pain assessed through visual analogue scale (VAS) rating 0(no pain) to 10(extreme pain) were given individually to participant to gather information. The lower the score, the lesser the pain and vise versa.

CONTACTS AND LOCATIONS:
Overall Officials: Chia Jung Lee, Principal Investigator — University Alfonso X El Sabio
Locations (1):
- Centro Odonologico Innovacion y Especilidades Avanzadas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data could be shared for further analysis or comparison to other researchers

REFERENCES:
- [Background] Scheurer PA, Firestone AR, Burgin WB. Perception of pain as a result of orthodontic treatment with fixed appliances. Eur J Orthod. 1996 Aug;18(4):349-57. doi: 10.1093/ejo/18.4.349. PMID 8921656
- [Background] Cardoso PC, Espinosa DG, Mecenas P, Flores-Mir C, Normando D. Pain level between clear aligners and fixed appliances: a systematic review. Prog Orthod. 2020 Jan 20;21(1):3. doi: 10.1186/s40510-019-0303-z. PMID 31956934
- [Background] Krukemeyer AM, Arruda AO, Inglehart MR. Pain and orthodontic treatment. Angle Orthod. 2009 Nov;79(6):1175-81. doi: 10.2319/121308-632R.1. PMID 19852612
- [Background] Banerjee S, Banerjee R, Shenoy U, Agarkar S, Bhattacharya S. Effect of orthodontic pain on quality of life of patients undergoing orthodontic treatment. Indian J Dent Res. 2018 Jan-Feb;29(1):4-9. doi: 10.4103/ijdr.IJDR_113_16. PMID 29442079
- [Background] Kafle D, Rajbhandari A. Anticipated pain and pain experience among orthodontic patients: is there any difference? Kathmandu Univ Med J (KUMJ). 2012 Apr-Jun;10(38):71-3. doi: 10.3126/kumj.v10i2.7348. PMID 23132480
- [Background] Nicotra C, Polizzi A, Zappala G, Leonida A, Indelicato F, Caccianiga G. A Comparative Assessment of Pain Caused by the Placement of Banded Orthodontic Appliances with and without Low-Level Laser Therapy: A Randomized Controlled Prospective Study. Dent J (Basel). 2020 Mar 4;8(1):24. doi: 10.3390/dj8010024. PMID 32143365
- See also: The Visual analogue Scale (VAS) for pain assessment — https://www.physio-pedia.com/Visual_Analogue_Scale
- See also: Questionnaire designed and distributed through this website — https://www.surveyhero.com

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04834466/Prot_000.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04834466/ICF_001.pdf